CLINICAL TRIAL: NCT02025049
Title: Pilot Trial of Intravenous DP-b99 in the Treatment of First-ever Episode of Non-obstructive Acute High-risk Pancreatitis
Brief Title: DP-b99 in the Treatment of Acute High-risk Pancreatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: D-Pharm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ptcl-01501
Record Dates: First submitted 2013-12-25; First posted 2013-12-31 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2013-12

CONDITIONS: Pancreatitis
Keywords: pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — DP-b99

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DP-b99 (Experimental): Intravenous DP-b99, 1.0 mg/kg twice daily for 2 consecutive days
  Interventions: Drug: DP-b99
- Placebo (Placebo Comparator): Intravenous placebo (mannitol based, DP-b99 look-alike) twice daily for 2 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DP-b99 — DP-b99 is a lipophilic analog of the divalent metal ion chelator O,O'-Bis(2-aminophenyl) ethyleneglycol-N,N,N',N'-tetraacetic acid (BAPTA)
  Other Names: Chemical name: 1,2-Bis(2-aminophenoxy)ethane- N,N,N'N'-tetraacetic acid, N,N'-di(octyloxyethyl ester), N,N'-disodium salt; CAS Number: 222315-66-4
  Arms: DP-b99
Drug: Placebo — mannitol-based DP-b99 look-alike
  Arms: Placebo

SUMMARY:
Inflammation of the pancreas often leads to severe damage not only to the pancreas but also to other organs in the abdomen as well as to complications in organs further away like the lung and the kidney. This trial will examine if DP-b99, given to patients with non-severe inflammation of the pancreas, can mitigate the development of processes that can lead to serious complications of this disease.

DETAILED DESCRIPTION:
The study will be a randomised, double blind, placebo-controlled, multi-centre, multi-national, parallel-arm study comparing a placebo group to a DP-b99 group treated intravenously with 1.0 mg/kg twice daily for 2 consecutive days.

The study will enrol 30 patients at high risk of developing severe pancreatitis, as assessed by the Bedside Index for Severity in Acute Pancreatitis (BISAP) score of 3 or more at study entry.

The primary study endpoint is the effect of DP-b99 on systemic inflammation in acute pancreatitis as reflected by C-reactive protein (CRP) plasma levels. The secondary endpoints are the safety of DP-b99 in this population of patients (through routine safety laboratory tests, physical examination and vital signs monitoring, ECG and adverse event reporting), DP-b99's effects on other plasma inflammatory markers (interleukin-6, matrix metalloproteinase 9, tumor necrosis factor alpha) as well as its effects on the clinical course of pancreatitis (based on changes in the Systemic Inflammatory Response Syndrome (SIRS) and Acute Physiology And Chronic Health Evaluation II (APACHE II) scores, and on contrast material-enhanced abdominal Computerised Tomography (CT), versus placebo.

Clinical trial material administration will begin within 48 hours of acute pancreatitis symptoms onset. Subjects will be randomised at a ratio of 1:1 to receive either DP b99 or placebo. The serum levels of DP-b99 at the end of each 2-hour infusion will also be monitored.

The study duration per individual subject will be 14 days, consisting of a screening evaluation followed by a 48-hour double blind treatment period, which will be part of an in-hospital observation period of at least 6 days, and a follow-up final visit on Day 14.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject.
* Age 18 years or higher.
* First in a lifetime episode of acute pancreatitis.
* Diagnosis of acute pancreatitis based on 2 of the following 3 criteria: (1) typical upper abdominal pain; (2) elevation of serum amylase and/or lipase at least 3 times the upper limit of normal; (3) contrast-material enhanced CT scan or abdominal sonogram demonstrating changes of acute pancreatitis
* History supporting alcoholic, hypertriglyceridemic or biliary etiology of the current pancreatitis episode (for biliary pancreatitis, a sonogram must exclude a stone obstruction at the time of study screening).
* BISAP score of 3 or higher
* Study treatment initiation is possible within 48 h of symptom onset
* Ability to provide informed consent

Exclusion Criteria:

* Drug-induced, viral, hereditary or post-ERCP pancreatitis.
* Recurrent episode of pancreatitis.
* CT evidence of pancreatic necrosis at study entry.
* Imaging evidence of physical obstruction of the common bile duct at study entry; e.g. for abdominal sonogram, stone(s) in the common bile duct or common bile duct having diameter less than 6 mm (above 80 years, less than 8 mm) with gallbladder in situ.
* Severe chronic renal failure (Modification of Diet in Renal Disease formula 30 mL/min or dependency on renal dialysis).
* High likelihood for an invasive intra-biliary tract intervention (e.g. ERCP) in the coming week.
* Class II or greater New York Heart Association heart failure.
* Oxygen-dependent chronic obstructive pulmonary disease (COPD).
* Cirrhosis of the liver.
* Severe anemia (hemoglobin less than 8 g/dL).
* Hematocrit below 35 % or above 45 % at study entry (fluids may be administered to correct the hematocrit before randomisation as long as study treatment starts within 48 hours of symptoms onset).
* Serum alanine aminotransferase above 250 IU/L at study entry.
* Clinical suspicion of ascending cholangitis at study entry.
* Active gastrointestinal bleeding.
* Current malignancy not in remission (other than basal cell carcinoma of skin).
* Altered mental status.
* Current breastfeeding or pregnancy.
* Female of childbearing potential (less than 2 years postmenopausal or not surgically sterilized) who is not willing to use adequate and effective birth control measures
* Known hypersensitivity to any component of the investigational product.
* Dependent relationship with the investigator or the sponsor.
* Participation in an investigational drug study during this clinical trial or within 30 days prior to start of this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
C-reactive protein serum concentration | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Rosenberg, MD, Study Director — D-Pharm Ltd.
Locations (1):
- The University Hospital Brno, Gastroenterology Clinic, Brno, Czechia